CLINICAL TRIAL: NCT02014454
Title: Safety and Efficacy of Propranolol Eye Drops in Newborns With Retinopathy of Premature (DROP-PROP)
Brief Title: Safety and Efficacy of Propranolol Eye Drops in Treating Retinopathy of Premature
Acronym: DROP-PROP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Luca Filippi, MD, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DROP-PROP
Record Dates: First submitted 2013-12-10; First posted 2013-12-18 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of prematurity; Propranolol; Eye drops; Newborns; Retinal angiogenesis; Retinal neovascularization
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propranolol eye drops (Experimental): All the enrolled preterm newborns will receive propranolol as ophthalmic solution (0,1%): 3 microdrops of 6 microliters (μL) propranolol solution (= 6 μg propranolol/microdrop) will be topically applied with a calibrated pipette, in each eye, three times daily (every 8 hours).The treatment will continue until the complete development of retinal vascularization, but no more than 60 days.
  The propranolol treatment will be always associated to the conventional approach adopted by the Early Treatment for Retinopathy of Prematurity Study (ETROP Cooperative Group.
  Interventions: Drug: Propranolol eye drops

INTERVENTIONS:
Drug: Propranolol eye drops — All the enrolled preterm newborns will receive propranolol as ophthalmic solution (0,1%): 3 microdrops of 6 microliters (μL) propranolol solution (= 6 μg propranolol/microdrop) will be topically applied with a calibrated pipette, in each eye, three times daily (every 8 hours).The treatment will continue until the complete development of retinal vascularisation, but no more than 60 days.
  The propranolol treatment will be always associated to the conventional approach adopted by the ETROP Cooperative Group.

SUMMARY:
The aim of the present study is to evaluate the safety and efficacy of propranolol eye drops in preterm newborns with a precocious stage of retinopathy of prematurity (ROP). Preterm newborns (gestational age 23-32 weeks) with a stage 2 ROP (zone II without plus) will receive propranolol eye drops treatment until retinal vascularization will be completed.

Propranolol concentrations will be measured on dried blood spots during the first 3 days of treatment and at the steady state. Cardiovascular and respiratory parameters will be continuously monitored. Blood samplings checking metabolic, renal and liver functions will be performed periodically, as well as cardiac function, in order to verify the treatment safety. Serial ophthalmological evaluations will be planned to monitor the efficacy of the treatment, the ROP progression and the possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns (gestational age 23-32 weeks) with stage 2 ROP, zone II without plus.
* A signed parental informed consent.

Exclusion Criteria:

* Newborns with heart failure;
* Newborns with congenital cardiovascular anomalies, except for persistent ductus arteriosus, patent foramen ovale and small ventricular septal defects;
* Newborns with recurrent bradycardia (heart rate < 90 beat per minute);
* Newborns with second or third degree atrioventricular block;
* Newborns with hypotension;
* Newborns with renal failure;
* Newborns with actual cerebral haemorrhage;
* Newborns with other diseases which contraindicate the use of beta-adrenoreceptor blockers.

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of progression from stage 2 ROP to more severe stage ROP (stage 2 or 3 with plus, stage 4 and stage 5) | participants will be followed for the duration of hospital stay, an expected average of 2 months
  Eye drop propranolol is considered to be effective in counteracting the progression of ROP if the treatment decreases the incidence rate of progression from stage 2 ROP to more severe stage ROP (stage 2 or 3 with plus) from actual 38% to 19% or less.
Plasma concentrations of propranolol at the steady state | 10th day of treatment
  To evaluate the safety of eye drop propranolol we consider the plasma propranolol concentrations at the steady state. In particular it should be always less than 20 ng/ml, which is the plasma concentration, at the steady state, reported after oral administration of propranolol in the PROP-ROP study

SECONDARY OUTCOMES:
Number of newborns who progress to Stage 3 without plus ROP | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who progress to Stage 4 or 5 ROP with total or partial retinal detachment | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who need laser treatment | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who need rescue treatment with bevacizumab | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who need vitrectomy | participants will be followed for the duration of hospital stay, an expected average of 2 months
Collection of adverse events due to eye drop propranolol treatment | participants will be followed for the duration of hospital stay, an expected average of 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Luca Filippi, MD, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (2):
- Italy (2):
  - Neonatal Intensive Care Unit, A. Meyer University Childrens' Hospital, Florence
  - Institute of Pediatrics and Neonatology, Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, University of Milan, Milan

REFERENCES:
- [Background] Filippi L, Cavallaro G, Bagnoli P, Dal Monte M, Fiorini P, Donzelli G, Tinelli F, Araimo G, Cristofori G, la Marca G, Della Bona ML, La Torre A, Fortunato P, Furlanetto S, Osnaghi S, Mosca F. Oral propranolol for retinopathy of prematurity: risks, safety concerns, and perspectives. J Pediatr. 2013 Dec;163(6):1570-1577.e6. doi: 10.1016/j.jpeds.2013.07.049. Epub 2013 Sep 18. PMID 24054431
- [Background] Dal Monte M, Casini G, la Marca G, Isacchi B, Filippi L, Bagnoli P. Eye drop propranolol administration promotes the recovery of oxygen-induced retinopathy in mice. Exp Eye Res. 2013 Jun;111:27-35. doi: 10.1016/j.exer.2013.03.013. Epub 2013 Mar 23. PMID 23528535
- [Background] Filippi L, Cavallaro G, Fiorini P, Malvagia S, Della Bona ML, Giocaliere E, Bagnoli P, Dal Monte M, Mosca F, Donzelli G, la Marca G. Propranolol concentrations after oral administration in term and preterm neonates. J Matern Fetal Neonatal Med. 2013 May;26(8):833-40. doi: 10.3109/14767058.2012.755169. Epub 2013 Jan 31. PMID 23205867
- [Background] Della Bona ML, Malvagia S, Villanelli F, Giocaliere E, Ombrone D, Funghini S, Filippi L, Cavallaro G, Bagnoli P, Guerrini R, la Marca G. A rapid liquid chromatography tandem mass spectrometry-based method for measuring propranolol on dried blood spots. J Pharm Biomed Anal. 2013 May 5;78-79:34-8. doi: 10.1016/j.jpba.2013.01.034. Epub 2013 Feb 4. PMID 23434527
- [Derived] Filippi L, Cavallaro G, Bagnoli P, Dal Monte M, Fiorini P, Berti E, Padrini L, Donzelli G, Araimo G, Cristofori G, Fumagalli M, la Marca G, Della Bona ML, Pasqualetti R, Fortunato P, Osnaghi S, Tomasini B, Vanni M, Calvani AM, Milani S, Cortinovis I, Pugi A, Agosti M, Mosca F. Propranolol 0.1% eye micro-drops in newborns with retinopathy of prematurity: a pilot clinical trial. Pediatr Res. 2017 Feb;81(2):307-314. doi: 10.1038/pr.2016.230. Epub 2016 Nov 4. PMID 27814346